CLINICAL TRIAL: NCT05119166
Title: International Milk Composition (IMiC) Consortium
Acronym: IMiC
Status: Active, not recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Stanford University (Other); The University of Western Australia (Other); University of Idaho (Other); Ludwig-Maximilians - University of Munich (Other); Johns Hopkins University (Other); Cedars-Sinai Medical Center (Other); Sapient Bioanalytics (Unknown); University of California, Davis (Other); University of California, San Diego (Other); University of Virginia (Other); Aga Khan University (Other); University Ghent (Other); University of California, Berkeley (Other); University Health Network, Toronto (Other); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency); Antigen Discovery Inc (Unknown); USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: HS23767; H2020:161 (Other: University of Manitoba)
Record Dates: First submitted 2021-11-01; First posted 2021-11-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Infant Growth; Maternal Health; Infant Nutrition
MeSH Terms: interventions — Niacinamide; Azithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human Breast Milk Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Canadian Healthy Infant Longitudinal Development (CHILD) Cohort Study: The CHILD Cohort Study is a prospective longitudinal birth cohort study. It is an observational study of healthy term infants in Canada (Vancouver, Edmonton, Manitoba, Toronto). The birth years were between 2009-2012, and is currently at the 8 year postnatal follow up phase. IMiC will receive 400 breast milk samples from 400 dyads (100/site) that were taken between 3-4 months postnatal.
- The Early Life Interventions for Childhood Growth and Development in Tanzania (ELICIT) Study: (NCT03268902). ELICIT is a randomized controlled trial (RCT) evaluating the efficacy of antimicrobials and nicotinamide in increasing growth in the setting of Rural Tanzania. It is factorial design RCT of nicotinamide (vitamin B3) to mothers and infants, and antimicrobial prophylaxis to infants. IMiC will receive 400 breast milk samples from 200 dyads, 2 samples per dyad taken at 1 & 5 months postnatal.
  Interventions: Dietary Supplement: Vitamin B3; Biological: Azithromycin
- VITAL Pakistan: Two Randomized Controlled Trials: Mumta (Nutritional support for lactating women with or without azithromycin)PW - NCT04012177 and MumtaLW - NCT03564652 VITAL is a community-based, randomized control, assessor blinded trial in peri-urban settings of Karachi, Pakistan to study the impact of Lipid-based Nutritional Supplement for Pregnant and Lactating women which is balanced energy-protein (BEP) dietary supplement, a locally produced ready-to-use nutritional product for lactating women (LW) and single prophylaxis dose of Azithromycin for infants, on growth of infants over the period of six months since birth compared to current standard of care. IMiC will receive 600 breast milk samples from 200 dyads, 3 samples per dyad taken at 0-1, 1-2 & 2-3 months.
  Interventions: Biological: Azithromycin; Dietary Supplement: Fortified food supplement
- Micronutriments pour la Santé de la Mère et de l'Enfant (MISAME)-3 study (NCT03533712): MISAME-3 is a randomized controlled clinical trial in the setting of Rural Burkina Faso. A BEP supplement provides less than 25% of protein of the total energy content, and includes different vitamins and minerals. The first part of an exploratory study will determine which type of BEP supplement (bar, drink, biscuit, soup or paste) is most accepted by pregnant women. Subsequently, two products will be tested for longer-term acceptability and at-home use (phase 1). The effect of the most suitable supplement will be tested in a controlled clinical trial (phase 2). The intervention group will receive the dietary supplement during pregnancy and/or lactation, while the control group complies with the standard iron and folic acid tablets following the national guidelines. IMiC will receive 600 breast milk samples from 200 dyads, 3 samples per dyad taken at 0-1, 1-2 & 3-4 months.
  Interventions: Dietary Supplement: Fortified food supplement

INTERVENTIONS:
Dietary Supplement: Vitamin B3 — ELICIT Study: Factorial design RCT of nicotinamide (vitamin B3) to mothers and infants, and antimicrobial prophylaxis (Azithromycin) to infants.
  Other Names: Nicotinamide
  Groups: The Early Life Interventions for Childhood Growth and Development in Tanzania (ELICIT) Study
Biological: Azithromycin — ELICIT Study: Factorial design RCT of nicotinamide (vitamin B3) to mothers and infants, and antimicrobial prophylaxis (Azithromycin) to infants.
  VITAL Pakistan Study: 3-arm RCT of fortified food supplement (protein energy) during lactation, with or without azithromycin prophylaxis for infant.
  Groups: The Early Life Interventions for Childhood Growth and Development in Tanzania (ELICIT) Study; VITAL Pakistan
Dietary Supplement: Fortified food supplement — VITAL Study: 3-arm RCT of fortified food supplement (protein energy) during lactation, with or without azithromycin prophylaxis for infant.
  MISAMEIII Study: 2x2 cross-over efficacy RCT of fortified food supplement (folic acid/iron +/- peanut spread) during pregnancy and/or lactation; unmasked (open label).
  Groups: Micronutriments pour la Santé de la Mère et de l'Enfant (MISAME)-3 study (NCT03533712); VITAL Pakistan

SUMMARY:
The IMiC Consortium will analyze milk from 1000 mother-infant dyads across 4 diverse settings (Tanzania, Pakistan, Burkina Faso and Canada). Samples will be stored centrally at the Manitoba Interdisciplinary Lactation Centre (MILC) biorepository and distributed to multiple laboratories for analysis of macronutrients, micronutrients, oligosaccharides, growth factors, immunoglobulins, cytokines, metabolites and microbes. Data will be harmonized and stored in a central database, and diverse statistical methods will be applied for data integration and analysis.

DETAILED DESCRIPTION:
Human Milk Composition: Milk is a highly complex biofluid that has evolved over millions of years to nourish infants and protect them from infection while their immune system matures. In addition to delivering complete nutrition (i.e. macronutrients and micronutrients), milk provides bioactive components that further support infant growth, development and health. These include immunoglobulins, antibodies, hormones, growth factors, prebiotic oligosaccharides, and probiotic bacteria. Milk composition is specifically adapted to each mammalian species depending on the growth requirements of their young offspring. For example, the average energy content of human milk is around 70 kcal/100g, compared to 38 kcal/100g in donkey milk and 171 kcal/100g in mouse milk. Mice produce just 2 milk oligosaccharides, while humans produce over 150. Even among humans, milk composition is highly variable - for example, energy content can range from 57-83 kcal/100g and oligosaccharide concentrations range from 5-25 g/L.

Surprisingly little is known about the determinants and consequences of this variation. The investigators will study the following milk components in the IMiC Consortium to understand variability between individual women and across different geographic settings, and their associations with infant growth. In addition, to guide these analyses, a review of human milk components and infant growth will be undertaken by the IMiC members during Year 1 of the Project.

Priority Components (to be analyzed in all samples):

Macronutrients include carbohydrates (primarily lactose), proteins and lipids. Lipids provide about 50% of the energy content in human milk. The vast majority (98%) of milk lipids are triacylglycerides, with the remainder consisting of diacylglycerides, monoacylglycerides, free fatty acids, phospholipids and cholesterol. The fatty acid profile of human milk varies in relation to maternal diet and genetics, particularly in the long-chain polyunsaturated fatty acids (LCPUFAs), such as arachidonic and docosahexaenoic acids, which contribute to immune function and neurodevelopment.

Micronutrient quality and concentrations can be compromised by maternal malnutrition. Micronutrients in milk include minerals (e.g. Zinc, Calcium, Phosphorus, Magnesium, Iodine, Selenium) and vitamins (A, B1, B2, B6, B12, C, D, E; folate, choline).

Immunoglobulins (Ig) are transferred in human milk, including IgA, IgM and IgG. Infants are born with immature adaptive immunity, and rely on these maternal antibodies for defense against pathogens. Soluble IgA (sIgA) is the predominant antibody of human milk; sIgA-antigen complexes are taken up by intestinal dendritic cells, allowing for antigen recognition.

Cytokines are multifunctional peptides can cross the intestinal barrier, where they influence immune activity. Milk-borne cytokines include anti-inflammatory transforming growth factor (TGF)-b, interleukins (IL)-10 and IL-7, and proinflammatory tumor necrosis factor (TNF)-a, IL-6, IL-8, and interferon (IFN)-g.

Lactoferrin is an iron binding glycoprotein with antimicrobial activity against many bacteria, viruses, and fungi. Osteopontin is an extensively phosphorylated acidic glycoprotein that is present at high concentrations in human milk. It affects immune functions, intestinal development, and brain development.

Growth factors and hormones in human milk have wide-ranging effects on the infant intestinal tract, vasculature, nervous system, and endocrine system. Some act locally on the neonatal intestine and many are absorbed into systemic circulation through the 'leaky' infant gut. Epidermal growth factor (EGF) is critical to the maturation and healing of the intestinal mucosa. Insulin-like growth factor (IGF) promotes tissue growth. The metabolic hormones leptin, insulin, adiponectin and ghrelin regulate energy conservation, appetite and infant BMI.

Human milk oligosaccharides (HMOs) are the third most abundant component of human milk. Over 100 different HMOs have been identified. These structurally diverse carbohydrates are not digested by the infant, but are metabolized by the infant's gut bacteria, providing a selective substrate to help shape the developing microbiome. In addition, HMOs serve as soluble decoy receptors and prevent pathogen attachment to infant mucosal surfaces, lowering the risk for viral and bacterial infections. HMOs may also modulate epithelial and immune cell responses and provide the infant with sialic acid, an important nutrient for brain development. In the CHILD cohort the investigators have observed that, beyond genetic secretor status, HMO composition is associated with ethnicity, lactation stage, parity, geographic location, season of collection, and breastfeeding exclusivity.

Omics approaches will be applied to broadly assess the complete spectrum of peptides, proteins, lipids, and metabolites in human milk. Targeted metabolomics analyses to be conducted using the Biocrates platform (~500 metabolites), untargeted metabolomic analyses to be conducted by Sapient Bioanalytics via mass spectrometry.

Microbes are present in human milk. Culture-dependent and independent (sequencing-based) studies have confirmed the presence of bacteria and fungi in milk from healthy mothers. In the CHILD cohort, the investigators have found that milk microbiota composition differs by infant sex, method of feeding, maternal BMI, and maternal atopy. It is estimated that breastfed infants receive 10^4-10^6 bacteria per day, providing a source of live microbes to seed the infant gut, oral cavity and airways. Studies demonstrating strain similarities between maternal gut, milk, and infant gut support this hypothesis, and find that Bifidobacterium spp. constitute the majority of shared taxa between maternal milk and infant stool. Given the central role of the gut microbiome in infant growth, metabolism and protection from infectious disease, including in low to middle income (LMIC) settings, it is critical to understand the origins of these fundamentally important gut microbes early in life.

A secondary objective of IMiC will be to support data integration across sites to answer important questions related to 1) the impact of maternal health and nutrition interventions on breast milk composition, and 2) its relation to infant health, growth and development. Each site will own its own data and will also be independently addressing these same questions by site, as originally intended in their own grants/studies.

ELIGIBILITY:
Inclusion Criteria:

* CHILD Study: Full term healthy infant; singleton pregnancy; English literary
* ELICIT Study: Adult mothers, child <14 days, lives within 25km of Haydom
* VITAL Study: Lactating, biological mothers
* MISAMEIII Study: Confirmed (pregnancy test/ultrasound) pregnant women 15-40 years old, informed consent, self, parents or husband (for minors; assent).

Exclusion Criteria:

* CHILD Study: IVF; congenital abnormality; preterm delivery
* ELICIT Study: Multiple gestation, birth defects/neonatal illness, weight <1.5g, no intention to breastfeed, will move from area within 18 months
* VITAL Study: Use of any ointments or topical solutions immediately prior to sampling, non-consent
* MISAMEIII Study: Peanut allergy, gestational age <20weeks, women who will not deliver babies in or live in study area by delivery date.

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: CHILD Study: observational study of healthy term infants from Canada, Multi-ethnic (~70% Caucasian; 30% others: Asian, First Nations, Black, other) ELICIT Study: factorial RCT study design, cohorts from Haydom, Tanzania, predominantly of Black and East African descent VITAL Study: 3-arm RCT study design, cohorts from Karachi, Pakistan, predominantly of Asian descent MISAMEIII Study: 2x2 cross-over RCT study design, cohorts from Hounde District, Burkina Faso, predominantly of Black and West African descent
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-17 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Create an international consortium of 4 birth cohorts in Tanzania, Pakistan, Burkina Faso and Canada (Field Site Partners), human milk scientists (Laboratory Partners), and data scientists and biostatisticians (Data Science Partners). | This outcome is anticipated to reach completion in December 2021.
  The result of this outcome will be measured by the completion of governance structure and data sharing agreements with all partners.
Create a centralized biorepository of human milk samples from the Field Site Partners, housed at the Manitoba Interdisciplinary Lactation Centre (MILC) at the University of Manitoba in Winnipeg, Manitoba, Canada. | This outcome is anticipated to reach completion in April 2022.
  The result of this outcome will be measured by the completion of all milk samples collected, stored and catalogued at MILC.
Create a standardized protocol for the comprehensive analysis of human milk composition using state-of-the-art methods in expert laboratories | This outcome is anticipated to reach completion in December 2021.
  The result of this outcome will be measured by the completion of list of target milk components; agreements with laboratories; standard operating procedures (SOPs) for sample collection, processing, shipping and analysis.
Create a harmonized dataset of human milk composition and relevant maternal, infant and environmental data from 1000 dyads | This outcome is anticipated to reach completion in October 2023.
  The result of this outcome will be measured by complete, clean, accessible, dataset meeting FAIR (Findable, Accessible, Interoperable, Reusable: www.gofair.org) Guiding Principles, including milk composition data and relevant metadata for all included dyads.
Create an integrated analysis of this dataset | This outcome is anticipated to reach completion in October 2023.
  Create an integrated analysis of this dataset, addressing research questions such as:
  * What are the ranges and distributions of analytes in human milk in different geographic settings?
  * How are various components in human milk correlated with each other?
  * How is breast milk composition influenced by maternal, environmental and sociodemographic factors? The result of this outcome will be measured by answering the above research questions, compiled in reports and open access academic publications

SECONDARY OUTCOMES:
A secondary objective of IMiC will be to support data integration across sites to answer important questions. | This outcome is anticipated to reach completion in October 2023.
  A secondary objective of IMiC will be to support data integration across sites to answer important questions related to 1) the impact of maternal health and nutrition interventions on breast milk composition, and 2) its relation to infant health, growth and development. Each site will own its own data and will also be independently addressing these same questions by site, as originally intended in their own grants/studies.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Azad, Principal Investigator — University of Manitoba, CHILD Cohort Study; Estomih Mduma, Study Director — Haydom Lutheran Hospital, ELICIT Trial; Fyezah Jehan, Principal Investigator — Aga Khan University Pakistan, VITAL Trial; Laeticia Celine Toe, Study Director — Institut de Recherche en Science de la Santa, MISAMEIII Trial; PJ Subbarao, Study Director — SickKids, CHILD Study; Yasir Shafiq, Principal Investigator — Aga Khan University Pakistan, VITAL Trial; Mark D DeBoer, Principal Investigator — University of Virginia, VITAL Trial; Patrick Kolsteren, Principal Investigator — Ghent University, MISAMEIII Trial
Locations (1):
- Manitoba Interdisciplinary Lactation Centre (MILC), Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared: final, annotated datasets and associated documentation (protocols, questionnaires, codebooks, data dictionaries, etc.). Data will be deposited into an open access data repository.
Supporting Information: Study Protocol, SAP
Time Frame: Embargo period of 12 months followed by full open access
Access Criteria: Embargo period of 12 months followed by full open access

REFERENCES:
- [Background] Andreas NJ, Kampmann B, Mehring Le-Doare K. Human breast milk: A review on its composition and bioactivity. Early Hum Dev. 2015 Nov;91(11):629-35. doi: 10.1016/j.earlhumdev.2015.08.013. Epub 2015 Sep 12. PMID 26375355
- [Background] Ballard O, Morrow AL. Human milk composition: nutrients and bioactive factors. Pediatr Clin North Am. 2013 Feb;60(1):49-74. doi: 10.1016/j.pcl.2012.10.002. PMID 23178060
- [Background] Bode L. Human milk oligosaccharides: every baby needs a sugar mama. Glycobiology. 2012 Sep;22(9):1147-62. doi: 10.1093/glycob/cws074. Epub 2012 Apr 18. PMID 22513036
- [Background] Azad MB, Robertson B, Atakora F, Becker AB, Subbarao P, Moraes TJ, Mandhane PJ, Turvey SE, Lefebvre DL, Sears MR, Bode L. Human Milk Oligosaccharide Concentrations Are Associated with Multiple Fixed and Modifiable Maternal Characteristics, Environmental Factors, and Feeding Practices. J Nutr. 2018 Nov 1;148(11):1733-1742. doi: 10.1093/jn/nxy175. PMID 30247646
- [Background] Innis SM. Impact of maternal diet on human milk composition and neurological development of infants. Am J Clin Nutr. 2014 Mar;99(3):734S-41S. doi: 10.3945/ajcn.113.072595. Epub 2014 Feb 5. PMID 24500153
- [Background] Dror DK, Allen LH. Overview of Nutrients in Human Milk. Adv Nutr. 2018 May 1;9(suppl_1):278S-294S. doi: 10.1093/advances/nmy022. PMID 29846526
- [Background] Dawod B, Marshall JS. Cytokines and Soluble Receptors in Breast Milk as Enhancers of Oral Tolerance Development. Front Immunol. 2019 Jan 22;10:16. doi: 10.3389/fimmu.2019.00016. eCollection 2019. PMID 30723472
- [Background] Garofalo R. Cytokines in human milk. J Pediatr. 2010 Feb;156(2 Suppl):S36-40. doi: 10.1016/j.jpeds.2009.11.019. PMID 20105664
- [Background] Demmelmair H, Prell C, Timby N, Lonnerdal B. Benefits of Lactoferrin, Osteopontin and Milk Fat Globule Membranes for Infants. Nutrients. 2017 Jul 28;9(8):817. doi: 10.3390/nu9080817. PMID 28788066
- [Background] Jiang R, Lonnerdal B. Biological roles of milk osteopontin. Curr Opin Clin Nutr Metab Care. 2016 May;19(3):214-9. PMID 27504516
- [Background] Chan D, Goruk S, Becker AB, Subbarao P, Mandhane PJ, Turvey SE, Lefebvre D, Sears MR, Field CJ, Azad MB. Adiponectin, leptin and insulin in breast milk: associations with maternal characteristics and infant body composition in the first year of life. Int J Obes (Lond). 2018 Jan;42(1):36-43. doi: 10.1038/ijo.2017.189. Epub 2017 Aug 14. PMID 28925410
- [Background] Young BE, Patinkin Z, Palmer C, de la Houssaye B, Barbour LA, Hernandez T, Friedman JE, Krebs NF. Human milk insulin is related to maternal plasma insulin and BMI: but other components of human milk do not differ by BMI. Eur J Clin Nutr. 2017 Sep;71(9):1094-1100. doi: 10.1038/ejcn.2017.75. Epub 2017 May 17. PMID 28513622
- [Background] Moossavi S, Miliku K, Sepehri S, Khafipour E, Azad MB. The Prebiotic and Probiotic Properties of Human Milk: Implications for Infant Immune Development and Pediatric Asthma. Front Pediatr. 2018 Jul 24;6:197. doi: 10.3389/fped.2018.00197. eCollection 2018. PMID 30140664
- [Background] Musilova S, Rada V, Vlkova E, Bunesova V. Beneficial effects of human milk oligosaccharides on gut microbiota. Benef Microbes. 2014 Sep;5(3):273-83. doi: 10.3920/BM2013.0080. PMID 24913838
- [Background] Wang B. Molecular mechanism underlying sialic acid as an essential nutrient for brain development and cognition. Adv Nutr. 2012 May 1;3(3):465S-72S. doi: 10.3945/an.112.001875. PMID 22585926
- [Background] McGuire MK, McGuire MA. Got bacteria? The astounding, yet not-so-surprising, microbiome of human milk. Curr Opin Biotechnol. 2017 Apr;44:63-68. doi: 10.1016/j.copbio.2016.11.013. Epub 2016 Dec 8. PMID 27940404
- [Background] Ruiz L, Garcia-Carral C, Rodriguez JM. Unfolding the Human Milk Microbiome Landscape in the Omics Era. Front Microbiol. 2019 Jun 25;10:1378. doi: 10.3389/fmicb.2019.01378. eCollection 2019. PMID 31293535
- [Background] Togo A, Dufour JC, Lagier JC, Dubourg G, Raoult D, Million M. Repertoire of human breast and milk microbiota: a systematic review. Future Microbiol. 2019 May;14:623-641. doi: 10.2217/fmb-2018-0317. Epub 2019 Apr 26. PMID 31025880
- [Background] Moossavi S, Sepehri S, Robertson B, Bode L, Goruk S, Field CJ, Lix LM, de Souza RJ, Becker AB, Mandhane PJ, Turvey SE, Subbarao P, Moraes TJ, Lefebvre DL, Sears MR, Khafipour E, Azad MB. Composition and Variation of the Human Milk Microbiota Are Influenced by Maternal and Early-Life Factors. Cell Host Microbe. 2019 Feb 13;25(2):324-335.e4. doi: 10.1016/j.chom.2019.01.011. PMID 30763539
- [Background] Asnicar F, Manara S, Zolfo M, Truong DT, Scholz M, Armanini F, Ferretti P, Gorfer V, Pedrotti A, Tett A, Segata N. Studying Vertical Microbiome Transmission from Mothers to Infants by Strain-Level Metagenomic Profiling. mSystems. 2017 Jan 17;2(1):e00164-16. doi: 10.1128/mSystems.00164-16. eCollection 2017 Jan-Feb. PMID 28144631
- [Background] Biagi E, Quercia S, Aceti A, Beghetti I, Rampelli S, Turroni S, Faldella G, Candela M, Brigidi P, Corvaglia L. The Bacterial Ecosystem of Mother's Milk and Infant's Mouth and Gut. Front Microbiol. 2017 Jun 30;8:1214. doi: 10.3389/fmicb.2017.01214. eCollection 2017. PMID 28713343
- [Background] Blanton LV, Barratt MJ, Charbonneau MR, Ahmed T, Gordon JI. Childhood undernutrition, the gut microbiota, and microbiota-directed therapeutics. Science. 2016 Jun 24;352(6293):1533. doi: 10.1126/science.aad9359. PMID 27339978
- [Background] Gehrig JL, Venkatesh S, Chang HW, Hibberd MC, Kung VL, Cheng J, Chen RY, Subramanian S, Cowardin CA, Meier MF, O'Donnell D, Talcott M, Spears LD, Semenkovich CF, Henrissat B, Giannone RJ, Hettich RL, Ilkayeva O, Muehlbauer M, Newgard CB, Sawyer C, Head RD, Rodionov DA, Arzamasov AA, Leyn SA, Osterman AL, Hossain MI, Islam M, Choudhury N, Sarker SA, Huq S, Mahmud I, Mostafa I, Mahfuz M, Barratt MJ, Ahmed T, Gordon JI. Effects of microbiota-directed foods in gnotobiotic animals and undernourished children. Science. 2019 Jul 12;365(6449):eaau4732. doi: 10.1126/science.aau4732. PMID 31296738
- [Background] Subramanian S, Huq S, Yatsunenko T, Haque R, Mahfuz M, Alam MA, Benezra A, DeStefano J, Meier MF, Muegge BD, Barratt MJ, VanArendonk LG, Zhang Q, Province MA, Petri WA Jr, Ahmed T, Gordon JI. Persistent gut microbiota immaturity in malnourished Bangladeshi children. Nature. 2014 Jun 19;510(7505):417-21. doi: 10.1038/nature13421. Epub 2014 Jun 4. PMID 24896187
- [Background] Foroutan A, Guo AC, Vazquez-Fresno R, Lipfert M, Zhang L, Zheng J, Badran H, Budinski Z, Mandal R, Ametaj BN, Wishart DS. Chemical Composition of Commercial Cow's Milk. J Agric Food Chem. 2019 May 1;67(17):4897-4914. doi: 10.1021/acs.jafc.9b00204. Epub 2019 Apr 17. PMID 30994344
- [Derived] Fehr K, Mertens A, Shu CH, Dailey-Chwalibog T, Shenhav L, Allen LH, Beggs MR, Bode L, Chooniedass R, DeBoer MD, Deng L, Espinosa C, Hampel D, Jahual A, Jehan F, Jain M, Kolsteren P, Kawle P, Lagerborg KA, Manus MB, Mataraso S, McDermid JM, Muhammad A, Peymani P, Pham M, Shahab-Ferdows S, Shafiq Y, Subramoney V, Sunko D, Toe LC, Turvey SE, Xue L, Rodriguez N, Hubbard A, Aghaeepour N, Azad MB. Protocol: the International Milk Composition (IMiC) Consortium - a harmonized secondary analysis of human milk from four studies. Front Nutr. 2025 Jun 10;12:1548739. doi: 10.3389/fnut.2025.1548739. eCollection 2025. PMID 40557242